CLINICAL TRIAL: NCT02936271
Title: Efficacy of Vasculera in Prevention on Post-op Pain and Edema Following Lower Extremity Venous Treatment in the Outpatient Setting.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-137
Record Dates: First submitted 2016-10-03; First posted 2016-10-18 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Venous Insufficiency of Leg; Venous Reflux; Varicose Veins; Lower Extremity Edema Chronic
Keywords: Radiofrequency Ablation; Sclerotherapy; Vasculera
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Vasculera (diosmiplex) (Active Comparator): Active Vasculera will be prescribed as one (1) tablet (630 mg) twice a day.
  Interventions: Other: Vasculera
- Vasculera Placebo (Placebo Comparator): Vasculera Placebo will be prescribed as one (1) tablet twice a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vasculera — Vasculera is a specially formulated prescription medical food product. This study compares Vasculera to placebo at reducing post procedural pain, bruising and edema for patients requiring an intervention for lower extremity venous disease.
  Patient will be randomized to receive Active Vasculera or Vasculera Placebo. The study product will be taken for two weeks prior to the patient's planned procedure and continued for four weeks after their procedure. If multiple procedures are required the patient will be instructed to use the product throughout treatment.
  Other Names: Diosmiplex; Prescription medical food product
  Arms: Active Vasculera (diosmiplex)
Other: Placebo
  Arms: Vasculera Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Vasculera in reducing post procedural pain, bruising and edema in the post procedure period for patients diagnosed with C2-C5 disease requiring an intervention(s).

The hypothesis is that Vasculera will reduce post procedural pain, bruising and edema for patients requiring an intervention.

This will be a randomized, double-blind, placebo-controlled study. Vasculera is a specially formulated prescription medical food product for the clinical dietary management of the metabolic processes of chronic venous insufficiency. Vasculera has limited side effects, please see the product insert.

A total of 110 patients will be enrolled into this study. Patients will be randomized to receive Vasculera (Study Product) or placebo. Study Product or placebo will be prescribed as one (1) tablet twice a day.

DETAILED DESCRIPTION:
Lower extremity venous disease is thought to affect 50 percent of woman and 40 percent of men at some point in their lifetime. Many of these patients seek venous treatment and undergo surgical procedures in the outpatient setting. Patient undergoing surgical intervention for treatment of venous reflux disease often experience discomfort, edema and discoloration in the areas of treatment. These symptoms may affect them for weeks to months after the procedure.

Radiofrequency ablation (RFA) of greater saphenous, small saphenous or accessory saphenous vein follow by sclerotherapy of remaining tributary veins 1-2 weeks later is a common minimally invasive treatment. Both the RFA and the ultrasound guided sclerotherapy cause an inflammatory response which can make the post-operative period more difficult for patients then the procedure itself.

Vasculara has been shown to reduce inflammation, improve vascular tone and decrease tissue acidosis. It has also been shown to be effective in the treatment of post phlebitic syndrome and may reduce thrombotic complication. Recent animal data has demonstrated decreased postsclerotherapy inflammation in rabbits. In anecdotal reports providers have had good result with prescribing this medication to patients to be take a week or two prior to the procedure and in the post-op period, however, evidence for this practice is lacking. Vasculara is a generally safe product with very limited side effects and thus could be applied to a large patient population if clear benefit were documented.

Vasculera is a prescription medical food product composed of the flavonoid, diosmin and a proprietary systemic blood alkalinizing agent, Alka4-complex. Diosmin has been used successfully in Europe for more than 35 years in the treatment of chronic venous insufficiency and its complications. There is a large body of published literature regarding the molecular activity, clinical efficacy and safety of diosmin as well as its effects on the microvasculature where it has been shown to reduce inflammation, improve structural integrity, improve capillary flow and reduce capillary leakage of serum proteins and red blood cells. It decreases bradykinin-induced microvascular leakage and may act favorably to inhibit leukocyte activation, trapping, and migration. Clinically, edema is reduced, ulcer healing is accelerated, and leukocyte trapping diminished.

A similar study with similar design to this study from a Russian group demonstrated the "feasibility of using the drug Detralex, a brand of diosmin marketed in Europe, as an agent for nonspecific pharmacological protection in endovascular treatment of varicose disease." In 2007 the DEFANS trial, also from Russia concluded, micronized diosmin in pre- and postoperative period after phlebectomy helps to attenuate pain syndrome, to decrease postoperative hematomas and accelerate their resorption, to increase exercise tolerance in early postoperative period. Studies performed within the United States with modern surgical procedures are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with C2-C5 disease undergoing radiofrequency ablation; foam and/or sclerotherapy
* Women of childbearing age must be using birth control to be candidates for study participation

Exclusion Criteria:

* Pregnant or nursing women
* Patients that are 85 years of age or older
* Patients who are unable to provide consent
* Prisoners or vulnerable population, including non-English speaking patients
* C1 Disease
* Patient on Chlorzoxazone, Diclofenac, Metronidazole
* Use of recreational drugs including alcohol in excess of 1 unit daily (for purposes of this study, a unit of alcohol is defined as 6 oz of wine, 12 oz of beer or 2 oz of hard spirits)
* Participation in another clinical trial within 7 half-lives of the prior study agent prior to the screening visit
* More than three planned surgical intervention procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Post-procedure Bruising | 2 weeks pre-procedure to 6 weeks post-procedure
  Physician and nurse examination
Post-procedure Bleeding | 2 weeks pre-procedure to 6 weeks post-procedure
  Physician and nurse examination
Post-procedure Pain | 2 weeks pre-procedure to 6 weeks post-procedure
  Pain scale
Post-procedure Edema | 2 weeks pre-procedure to 6 weeks post-procedure
  Physician and nurse examination

SECONDARY OUTCOMES:
Adverse Events | 2 weeks pre-procedure to 6 weeks post-procedure
  Adverse events per package insert.
Serious Adverse Events | 2 weeks pre-procedure to 6 weeks post-procedure
  Deep Vein Thrombosis (DVT) Pulmonary Embolism (PE) and Infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J. Watson, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brand FN, Dannenberg AL, Abbott RD, Kannel WB. The epidemiology of varicose veins: the Framingham Study. Am J Prev Med. 1988 Mar-Apr;4(2):96-101. PMID 3395496
- [Background] Callam MJ. Epidemiology of varicose veins. Br J Surg. 1994 Feb;81(2):167-73. doi: 10.1002/bjs.1800810204. PMID 8156326
- [Background] Zahariev T, Anastassov V, Girov K, Goranova E, Grozdinski L, Kniajev V, Stankev M. Prevalence of primary chronic venous disease: the Bulgarian experience. Int Angiol. 2009 Aug;28(4):303-10. PMID 19648874
- [Background] Bergan JJ. Chronic venous insufficiency and the therapeutic effects of Daflon 500 mg. Angiology. 2005 Sep-Oct;56 Suppl 1:S21-4. doi: 10.1177/00033197050560i104. PMID 16193222
- [Background] Tsimoyiannis EC, Floras G, Antoniou N, Papanikolaou N, Siakas P, Tassis A. Low-molecular-weight heparins and Daflon for prevention of postoperative thromboembolism. World J Surg. 1996 Oct;20(8):968-71; discussion 972. doi: 10.1007/s002689900145. PMID 8798349
- [Background] de Souza Md, Cyrino FZ, Mayall MR, Virgini-Magalhaes CE, Sicuro FL, de Carvalho JJ, Verbeuren TJ, Bouskela E. Beneficial effects of the micronized purified flavonoid fraction (MPFF, Daflon(R) 500 mg) on microvascular damage elicited by sclerotherapy. Phlebology. 2016 Feb;31(1):50-6. doi: 10.1177/0268355514564414. Epub 2014 Dec 15. PMID 25514922
- [Background] Lyseng-Williamson KA, Perry CM. Micronised purified flavonoid fraction: a review of its use in chronic venous insufficiency, venous ulcers and haemorrhoids. Drugs. 2003;63(1):71-100. doi: 10.2165/00003495-200363010-00005. PMID 12487623
- [Background] Ramelet AA. Clinical benefits of Daflon 500 mg in the most severe stages of chronic venous insufficiency. Angiology. 2001 Aug;52 Suppl 1:S49-56. doi: 10.1177/0003319701052001S07. PMID 11510597
- [Background] Shoab SS, Scurr JH, Coleridge-Smith PD. Plasma VEGF as a marker of therapy in patients with chronic venous disease treated with oral micronised flavonoid fraction - a pilot study. Eur J Vasc Endovasc Surg. 1999 Oct;18(4):334-8. doi: 10.1053/ejvs.1999.0890. PMID 10550269
- [Background] Bogachev VIu, Golovanova OV, Kuzhetsov AN, Shekoian AO. [On advisability of perioperative phleboprotection in endovascular treatment of lower in varicose disease: first initial results of the decision study]. Angiol Sosud Khir. 2012;18(2):90-5. Russian. PMID 22929677
- [Background] International Task Force. The management of chronic venous disorders of the leg: an evidence-based report of an international task force. Epidemiology. Phlebology. 1999;14(suppl 1):23-34.
- See also: Product website — http://www.vasculera.com/